CLINICAL TRIAL: NCT06564701
Title: A Pediatric Comparison of Remote Microphone Technologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: Hearts for Hearing (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SRF-22936
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-08

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Speech intelligibility testing will be conducted on a single group of participants, first using one remote mic system, and then the other. The order of devices will be counter-balanced across participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lab and Home Trial (Experimental): Participants who complete the lab testing, and who are able to use both devices during a field trial period in school
  Interventions: Device: Phonak Roger TouchScreen Microphone; Device: Phonak Partner Mic
- Experimental No Field Trial (Experimental): Participants who are only able to complete the lab testing
  Interventions: Device: Phonak Roger TouchScreen Microphone; Device: Phonak Partner Mic

INTERVENTIONS:
Device: Phonak Roger TouchScreen Microphone — Transmitter microphone system operating on the 2.4 GHz band, which allows for low-delay and reliable long-range broadcast to a compatible Roger receiver, designed to be used in educational settings. It features six microphones and adaptive technology in which speech signals are increased when background noise increases to ensure that the speech signal is always above the noise level.
Device: Phonak Partner Mic — Wireless microphone that uses Phonak proprietary AirStream technology to connect to Phonak hearing aids. It uses a fixed directional microphone, and is paired to the hearing aids such that the hearing aid microphones are attenuated at a fixed level when the microphone is in use.

SUMMARY:
Speech intelligibility will be evaluated for school age children with hearing loss in a simulated classroom environment, using Phonak hearing aids and receivers and two different microphone transmitters: a Roger Touchscreen mic and a fixed directional microphone.

DETAILED DESCRIPTION:
Speech intelligibility will be evaluated for school age children with hearing loss in a simulated classroom environment, using Phonak hearing aids and receivers and two different microphone transmitters: a Roger Touchscreen mic and a fixed directional microphone. The simulated classroom environment will include a teacher condition, in which speech is presented from a distance in front of the participant, and a small-group condition, in which speech is presented randomly from three different speakers around the participant. Both conditions will have diffuse background noise, and the various SNR (Signal to Noise Ratio) levels will be tested.

Subjective preference and fatigue questionnaires will also be collected from the participants after the use of each transmitter.

ELIGIBILITY:
Inclusion Criteria:

* Healthy middle and outer ear
* Mild, moderate or moderate-severe binaural sensorineural hearing loss
* Minimum AZ Bio score of 70% at 60 dB in quiet
* Experienced hearing aid users (6+ months)
* Able to read and follow directions
* English speakers with ability to communicate easily

Exclusion Criteria:

* Active middle ear infection
* Temporary or unilateral hearing loss
* Unable to follow verbal directions
* Unable to communicate easily
* Unable to tolerate the physical fit of the hearing aids

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
Speech Intelligibility score using the AZ Bio Sentence Test-teacher condition | One day (Visit 1)
  Sentences are presented from a front speaker located 8.5 feet away from participant. Diffuse background noise is presented from four corner speakers. Various Signal to Noise Ratios (SNR) will be tested: +4 dB, +2 dB, and -2 dB. The number of words correctly repeated will be calculated and expressed as a percentage for each SNR level. A higher score is better.
Speech Intelligibility score using the AZ Bio Sentence Test- small group condition | One day (Visit 1)
  Sentences are presented randomly from three different speakers, located around a small table with the participant, simulating a small group at a table. Diffuse background noise is presented from four corner speakers. Various Signal to Noise Ratios (SNR) will be tested: +4 dB, +2 dB, and -2 dB. The number of words correctly repeated will be calculated and expressed as a percentage for each SNR level. A higher score is better.

SECONDARY OUTCOMES:
Listening Fatigue using the Vanderbilt Fatigue Scale for Children | Two days (Visit 2 and Visit 3)
  Ten questions related to fatigue, answers rank from 1 (never) to 5 (almost always). Total scores can range from 10 to 50, with higher scores indicating more self-perceived fatigue.
Subjective Preferences of participants | Two days (Visit 1 following the lab testing, and Visit 3, following the field trial)
  Participants will be asked to rank their preference for the microphone systems using a Likert type of rating scale (1-5), where a lower score (<3) would indicate preference for the partner mic and a higher score (>3) will indicate preference for the Roger Touchscreen.

CONTACTS AND LOCATIONS:
Locations (1):
- Hearts for Hearing, Oklahoma City, Oklahoma, United States